CLINICAL TRIAL: NCT03738865
Title: G-Pen (Glucagon Injection) Compared to GlucaGen® Hypokit® (Glucagon) for Induced Hypoglycemia Rescue in Adults With T1D: A Phase 3 Multi-center, Randomized, Controlled, Single Blind, 2-way Crossover Study to Evaluate Efficacy and Safety
Brief Title: G-Pen Compared to Glucagen Hypokit for Severe Hypoglycemia Rescue in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: Empiristat, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XSGP-304
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Insulin Hypoglycemia; Type 1 Diabetes Mellitus; Severe Hypoglycemia
Keywords: glucagon; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G-Pen followed by Novo Glucagon (Experimental): 1 mg G-Pen at the first treatment visit followed by 1 mg Novo Glucagon at the second treatment visit
  Interventions: Drug: G-Pen; Drug: Novo Glucagon
- Novo Glucagon followed by G-Pen (Active Comparator): 1 mg Novo Glucagon at the first treatment visit followed by 1 mg G-Pen at the second treatment visit
  Interventions: Drug: G-Pen; Drug: Novo Glucagon

INTERVENTIONS:
Drug: G-Pen — 1 mg subcutaneous injection of G-Pen (glucagon injection) administered via auto-injector
  Other Names: glucagon
Drug: Novo Glucagon — 1 mg subcutaneous injection of Novo Glucagon (glucagon injection)
  Other Names: Glucagen Hypokit

SUMMARY:
This is a multi-center, randomized, controlled, single-blind, two-way crossover efficacy and safety study in subjects with Type 1 diabetes mellitus. The study involves two daytime clinical research center (CRC) visits with random assignment to receive G-Pen glucagon 1 mg during one period and Novo Glucagon 1 mg during the other. Each daytime visit is preceded by an overnight stay in the CRC. In the morning of the inpatient study visit, the subject is brought into a state of severe hypoglycemia through IV administration of regular insulin diluted in normal saline. After a hypoglycemic state with plasma glucose < 54 mg/dL (3 mmol/L) is verified, the subject is administered a dose of G-Pen or Novo Glucagon via subcutaneous injection. Plasma glucose levels are monitored for up to 180 minutes post-dosing, with a value of >70.0 mg/dL (3.89 mmol/L) or an increase of > 20 mg/dL (>1.11 mmol/L) within 30 minutes of glucagon administration indicating a positive response. After 3 hours, the subject is given a meal and discharged when medically stable. After a wash-out period of 7 to 28 days, subjects return to the CRC, and the procedures are repeated with each subject crossed over to the other treatment. A follow-up visit as a safety check is conducted 2-7 days following administration of the final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females diagnosed with type 1 diabetes (T1D) for at least 24 months.
2. Current usage of daily insulin treatment that includes having an assigned "correction factor" for managing hyperglycemia.
3. Age 18 to 75 years, inclusive.
4. Random serum C-peptide concentration < 0.6 ng/mL.
5. Willingness to follow all study procedures, including attending all clinic visits.
6. Subject has provided informed consent as evidenced by a signed and dated informed consent form (ICF) completed before any trial-related activities occur.

Exclusion Criteria:

1. Pregnancy
2. Glycated hemoglobin (HbA1c) > 10% at Screening.
3. Body mass index (BMI) > 40 kg/m2.
4. Renal insufficiency (serum creatinine greater than 3.0 mg/dL) or end-stage renal disease requiring renal replacement therapy.
5. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal to or greater than 3 times the upper limit of normal.
6. Hepatic synthetic insufficiency as defined as a serum albumin of less than 3.0 g/dL.
7. Hematocrit < 30%.
8. Blood pressure (BP) readings at Screening where systolic blood pressure (SBP) < 90 or > 150 mm Hg, and diastolic blood pressure (DBP) < 50 or > 100 mm Hg.
9. Clinically significant electrocardiogram (ECG) abnormalities.
10. Use of total insulin dose per day > 2 U/kg.
11. Inadequate venous access.
12. Congestive heart failure, New York Heart Association (NYHA) class III or IV.
13. History of myocardial infarction, unstable angina, or revascularization within the past 6 months.
14. History of a cerebrovascular accident in the past 6 months or with major neurological deficits.
15. Active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. Any history of breast cancer or malignant melanoma will be exclusionary.
16. Major surgical operation within 30 days prior to Screening.
17. Current seizure disorder (other than with suspect or documented hypoglycemia).
18. Current bleeding disorder, treatment with warfarin, or platelet count below 50 × 109 per liter.
19. History of pheochromocytoma or disorder with increased risk of pheochromocytoma (multiple endocrine neoplasia type 2 (MEN 2), neurofibromatosis, or Von Hippel-Lindau disease).
20. History of insulinoma.
21. History of allergies to glucagon or glucagon-like products, or any history of significant hypersensitivity to glucagon or any related products or to any of the excipients (DMSO and trehalose) in the investigational formulation.
22. History of glycogen storage disease.
23. Subject tests positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infection (hepatitis B surface antigen positive [HBsAg+]) at Screening.
24. Active substance other than tetrahydrocannabinol (THC) or alcohol abuse (more than 21 drinks per week for male subjects or 14 drinks per week for female subject).
25. Administration of glucagon within 7 days of Screening.
26. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before Screening for the current study and during participation in the current study.
27. Any other reason the Investigator deems exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - PPD-Las Vegas Clinical Research Unit, Las Vegas, Nevada
  - Rainier Research Center, Renton, Washington
- Medizinische Universität Graz-Center for Medical Research, Graz, Austria
- Canada (2):
  - LMC Diabetes & Endocrinology, Toronto, Ontario
  - AltaSciences, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieber TR, Aronson R, Christiansen MP, Bode B, Junaidi K, Conoscenti V. Efficacy, safety, tolerability, and noninferiority phase 3 study of glucagon as a ready-to-use room temperature liquid stable formulation versus a lyophilised formulation for the biochemical recovery and symptomatic relief of insulin-induced severe hypoglycaemia in adults with type 1 diabetes. Diabetes Obes Metab. 2022 Jul;24(7):1394-1397. doi: 10.1111/dom.14699. Epub 2022 Apr 28. No abstract available. PMID 35322535

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 132 subjects were randomized, however 1 subject withdrew prior to dosing, therefore 131 subjects received study drug.
Groups:
- G-Pen, Then Novo Glucagon: Participants first received G-Pen 1 mg subcutaneous injection each. After a washout period of 7-28 days, they then received Novo Glucagon 1 mg subcutaneous injection
- Novo Glucagon, Then G-Pen: Participants first received Novo Glucagon 1 mg subcutaneous injection each. After a washout period of 7-28 days, they then received G-Pen 1 mg subcutaneous injection
Period: Overall Study
Arm/Group | G-Pen, Then Novo Glucagon | Novo Glucagon, Then G-Pen
Started | 66 | 66
Completed | 61 | 62
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | G-Pen, Then Novo Glucagon | Novo Glucagon, Then G-Pen | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 63 | 126
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 37 | 33 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 65 | 63 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 2 | 2
  White | 62 | 61 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Severe Hypoglycemia Rescue
Description: Number of subjects with an increase in plasma glucose concentration from below 54 mg/dL (3 mmol/L) to greater than 70 mg/dL (3.89 mmol/L) or an increase in plasma glucose concentration > 20 mg/dL (> 1.11 mmol/L) within 30 minutes after administration of glucagon
Time Frame: At 30 minutes following administration of study drug
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- G-Pen: Participants received G-Pen 1 mg subcutaneous injection each.
- Novo Glucagon: Participants received Novo Glucagon 1 mg subcutaneous injection each.
Arm/Group | G-Pen | Novo Glucagon
Number analyzed (Participants) | 128 | 123
Participants | 127 | 123

2. Secondary Outcome: Plasma Glucose Response 1
Description: Number of subjects with an increase in plasma glucose concentration from below 54 mg/dL (3 mmol/L) to greater than 70 mg/dL (3.89 mmol/L) within 30 minutes of a decision to dose
Time Frame: At 30 minutes following a decision to administer study drug
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Novo Glucagon
Number analyzed (Participants) | 128 | 123
Participants | 127 | 123

3. Secondary Outcome: Plasma Glucose Response 2
Description: Number of subjects with an increase in plasma glucose concentration > 20 mg/dL (> 1.11 mmol/L) after administration of glucagon.
Time Frame: At 0-30 minutes following a decision to administer study drug
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Novo Glucagon
Number analyzed (Participants) | 128 | 123
Participants | 127 | 123

4. Secondary Outcome: Administration Time
Description: Mean time (minutes) to administer study drug from a decision to dose
Time Frame: At 0-10 minutes from a decision to administer study drug
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Novo Glucagon
Number analyzed (Participants) | 128 | 123
minutes | 0.79 (0.530) | 1.76 (0.678)

5. Secondary Outcome: Hypoglycemia Resolution
Description: Mean time (minutes) to complete resolution of the overall sensation of hypoglycemia from a decision to dose
Time Frame: At 0-90 minutes following administration of study drug
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Novo Glucagon
Number analyzed (Participants) | 128 | 123
minutes | 15.69 (7.428) | 15.32 (8.479)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 5 weeks, from the time of consent through the follow-up visit.
Description: Treatment-Emergent Adverse Events (TEAE) Note: Some subjects experienced multiple adverse events. Consequently, the sum of the number of subjects experiencing each individual adverse events is greater than the number of unique subjects experiencing at least one adverse event
Arm/Group | G-Pen | Novo Glucagon
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/123
Other Adverse Events (participants affected / at risk) | 67/127 | 57/123
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | G-Pen (N=127) | Novo Glucagon (N=123)
Nausea (Gastrointestinal disorders) | 54 | 55
Vomiting (Gastrointestinal disorders) | 16 | 17
Headache (Nervous system disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the Institution nor the principal investigator may submit for publication or presentation, the results of this trial without prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT03738865/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03738865/SAP_001.pdf